CLINICAL TRIAL: NCT04295681
Title: A Multicenter, Double-blind, Randomized, Parallel Group Placebo-controlled Clinical Trial of Efficacy and Safety of MMH-MAP in the Treatment of Cognitive Disorders in Patients With Ischemic Stroke in the Carotid Arteries
Brief Title: Clinical Trial of Efficacy and Safety of MMH-MAP in the Treatment of Cognitive Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-MAP-002
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMH-MAP (Experimental): Oral administration. 2 tablets twice daily (approximately at the same time). The drug is taken outside a meal (between the meals or 15 min prior to meal or fluid intake). Tablets should be held in the mouth until completely dissolved. The overall duration of treatment is 90 days.
  Interventions: Drug: MMH-MAP
- Placebo (Placebo Comparator): Oral administration. For 90 days according to MMH-MAP dosing regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MMH-MAP — Oral administration
  Other Names: Prospekta
  Arms: MMH-MAP
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The clinical trial to valuate efficacy and safety of MMH-MAP in the treatment of cognitive disorders in patients with ischemic stroke in the carotid arteries.

DETAILED DESCRIPTION:
Design: double-blind, randomized, parallel group placebo-controlled clinical study of efficacy and safety of MMH-MAP in the treatment of cognitive disorders in patients with ischemic stroke in the carotid arteries.

The study will enroll hospitalized subjects of either gender aged 40-75 years old with verified diagnosis of ischemic stroke in the carotid arteries within 72 hours post debut having moderate cognitive disorders, moderate neurological deficit.

At Visit 1 (day 1) the subject's complaints and medical history will be collected, objective examination, safety laboratory tests (hematology, serum chemistry, urinalysis) will be performed. The investigator will evaluate the patient's level of consciousness using The Glasgow Coma Scale, intensity of cognitive disorders using The Montreal Cognitive Assessment (МоСА), condition using National Institute of Health Stroke Scale (NIHSS) and The Modified Rankin Scale (mRs). Concomitant therapy will be recorded and changes in cerebral CT/MRI will be evaluated. If the subject meets inclusion criteria and has no exclusion criteria, he/she will be randomized to MMH-MAP or Placebo group. The first dose of the study product should be taken within 72 hours post stroke debut.

At Visit 2 (day 12±3, end of hospitalization period - the last day of hospitalization due to the current stroke) complaints will be collected, objective examination findings will be recorded, monitoring of the prescribed and concomitant therapy will be performed, treatment safety, compliance and stroke severity according to NIHSS will be evaluated.

By the end of hospital therapy the subject will be switched to outpatient therapy with continuation of IMP and medical assistance designed for the treatment of stroke and its sequelae.

At Visit 3 (day 45±7 days) the investigator will make a phone call to the subject evaluating the treatment safety.

At final Visit 4 (day 90±7 days) complaints will be collected, objective examination findings will be recorded, monitoring of the prescribed and concomitant therapy will be performed, treatment safety, compliance, condition according to NIHSS will be evaluated, mRs, Clinical Global Impression Efficacy Index (CGI-EI) will be filled. The investigator will perform MoCA testing. Safety laboratory tests (hematology, serum chemistry, urinalysis) will be carried out.

Throughout the study the patient will receive the treatment approved by the decree of the RF Ministry of Health dated 29.12.2012 No. 740n "On approval of standard of special care in cerebral infarction" except for the products specified in section "Forbidden concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years old inclusively.
2. Ischemic stroke in the carotid arteries (I 63) within 72 hours post debut.
3. Moderate cognitive disorders (MoCA < 26).
4. Normal consciousness (Glasgow score 15)
5. Stroke severity 8-12 according to NIHSS.
6. Disability mRs score 2-3.
7. Availability of cerebral CT/MRI within 72 hours post stroke debut.
8. Patients who agreed to use a reliable method of contraception during the study.
9. Patients who have signed the Participant Information Sheet and Informed Consent.

Exclusion Criteria:

1. Current or previous subarachnoidal/parenchymatous/ventricular hemorrhage, cerebral infarction, cerebral tumour.
2. Cerebral CT/MRI findings suggesting cerebral hemorrhage, tumour within 72 hours post stroke debut.
3. Scheduled or completed thrombolytic therapy for the treatment of the current cerebral infarction.
4. Central nervous system (CNS) diseases including:

   * Inflammatory diseases of the central nervous system (G00-G09);
   * Systemic atrophies primarily affecting the central nervous system (G10-G13);
   * Extrapyramidal and movement disorders (G20-G26);
   * Other degenerative diseases of the nervous system (G30-G32);
   * Demyelinating diseases of the CNS (G35-G37);
   * Episodic and paroxysmal disorders (G40-G47);
   * Polyneuropathies and other disorders of the peripheral nervous system (G60-64), with marked movement and/or sensory impairments that cause movement disorders;
   * Hydrocephalus (G91).
5. Head injuries (S00-S09) (including history), accompanied by impaired consciousness, brain contusion or open craniocerebral injuries.
6. Musculoskeletal disorders causing motor disturbances.
7. Dementia (including history) (F00-F03).
8. Malignant neoplasms.
9. Patients previously diagnosed with class IV heart failure (1964 New York Heart Association functional classification), hypothyroidism, or poorly treated diabetes mellitus.
10. Patients having unstable angina or myocardial infarction in the past 6 months.
11. Allergy/ intolerance to any of the components of medications used in the treatment.
12. Malabsorption syndrome, including congenital or acquired lactase deficiency (or any other disaccharidase deficiency) and galactosemia.
13. Any conditions which, according to the investigator opinion, may interfere with the subject's participation in the study.
14. Prior history of non-adherence to a drug regimen, a psychiatric disorder, alcoholism or drug abuse, which, in the opinion of the investigator, can compromise compliance with study protocol.
15. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial.
16. Participation in other clinical studies within 3 month prior to enrollment in the study.
17. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
18. Patients who work for OOO "NPF "Materia Medica Holding" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Russia (22):
  - The First City Clinical Hospital named after E.E. Volosevich, Arkhangelsk
  - Arkhangelsk Regional Clinical Hospital/Neurological Department, Arkhangelsk
  - Belgorod Regional Clinical Hospital of St. Joasaph, Belgorod
  - Regional Clinical Hospital # 3, Chelyabinsk
  - Kazan State Medical University/Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - Interregional Clinical Diagnostic Center, Kazan'
  - City Clinical Hospital # 7, Kazan'
  - Research Institute - Regional Clinical Hospital # 1 named after Prof. S.V. Ochapovsky, Krasnodar
  - City Clinical Hospital named after V.M. Buyanov, Moscow Department of Health, Moscow
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - City Clinical Hospital # 5 of the Nizhegorodskiy District of Nizhny Novgorod, Nizhny Novgorod
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Regional Clinic Hospital/Emergency cardiology unit with intensive care and resuscitation unit, Ryazan
  - St. Petersburg Research Institute of Ambulance named after I.I. Janelidze, Saint Petersburg
  - City Multidisciplinary Hospital # 2, Saint Petersburg
  - Samara City Clinical Hospital # 1 named after N.I. Pirogov/Neurological Department, Samara
  - Saratov City Clinical Hospital # 9, Saratov
  - Ulyanovsk Regional Clinical Hospital/Neurological Department, Ulyanovsk
  - Regional Clinic Hospital/Neurological department for patients with acute cerebrovascular accident, Vladimir
  - Voronezh Regional Clinical Hospital # 1, Voronezh
  - Vsevolozhsk Clinical Interdistrict Hospital, Vsevolozhsk
  - Clinical Hospital # 8/Intensive Care Unit, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 246 patients signed informed consent, of which 1 patient was excluded at the screening due to the patient's refusal to complete the MoCA scale.
Period: Overall Study
Arm/Group | MMH-MAP | Placebo
Started | 123 | 122
Completed | 122 | 119
Not Completed | 1 | 3
Not completed — Eligibility error | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMH-MAP | Placebo | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 63 | 129
  >=65 years | 57 | 59 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.4) | 62.5 (7.9) | 63.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 33 | 82
  Male | 74 | 89 | 163
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 123 | 122 | 245

OUTCOME MEASURES:

1. Primary Outcome: Average MoCA Score.
Description: Montreal Cognitive Assessment Scale (The Montreal Cognitive Assessment, MoCA) will be used to identify moderate cognitive impairment, as well as to assess changes in cognitive functions during therapy. The maximum possible number of points is 30; 26 points or more is considered normal. The minimum score is 0, higher score is better.
Time Frame: On baseline and on 90th day of the treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 122 | 119
score on a scale
  Baseline | 20.7 (3.5) | 21.7 (2.4)
  On 90th day of the treatment | 24.6 (2.9) | 24.5 (3.0)
  "90th day of the treatment minus baseline" score difference | 3.9 (2.5) | 2.9 (2.3)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Mean changes of MoCA scores (90th day of treatment minus baseline) were compared; Test type: Superiority; p = 0.0006, t-test, 2 sided; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [0.47 to 1.70] — Estimated value is calculated as "MMH-MAP minus Placebo" difference in mean MoCA scores changes

2. Secondary Outcome: Changes in NIHSS Score.
Description: NIHSS Scale (National Institutes of Health Stroke Scale) is a scale for assessing the severity of neurological disorders of the acute period of ischemic stroke. The NIHSS scale involves the assessment of a neurological condition by generally accepted methods of clinical examination of reflexes, sensory organs, and the patient's level of consciousness. The results range from minimum indicators - normal or close to normal, to maximum - reflect the degree of neurological damage. The score varies between 0 and 42, lower score is better.
Time Frame: On baseline, on 12th and on 90th days of the treatment.
Population: The number of completed cases (non-missing data) is indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 122 | 119
score on a scale
  Baseline | 8.6 (0.8) | 8.5 (0.7)
  On 12th day of the treatment: number analyzed (Participants) | 117 | 111
  On 12th day of the treatment | 4.9 (2.0) | 4.8 (1.9)
  On 90th day of the treatment: number analyzed (Participants) | 114 | 107
  On 90th day of the treatment | 3.0 (1.8) | 2.9 (1.8)
  "Baseline minus 12th day" score difference: number analyzed (Participants) | 117 | 111
  "Baseline minus 12th day" score difference | 3.6 (1.7) | 3.7 (1.9)
  "Baseline minus 90th day" score difference: number analyzed (Participants) | 114 | 107
  "Baseline minus 90th day" score difference | 5.6 (1.7) | 5.6 (2.0)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Mean changes of NIHSS scores (baseline minus 12th day of treatment) were compared; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.58 to 0.37] — Estimated value is calculated as "MMH-MAP minus Placebo" difference in mean MoCA scores changes
Statistical Analysis 2: Comparison: MMH-MAP vs Placebo; Mean changes of NIHSS scores (baseline minus 90th day of treatment) were compared; Test type: Superiority; p = 0.94, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.47 to 0.50] — Estimated value is calculated as "MMH-MAP minus Placebo" difference in mean MoCA scores changes

3. Secondary Outcome: Percentage of Patients With no Significant Disabilities.
Description: The modified Rankin scale (mRs 0-1) allows to assess the grade of disability after a stroke. The scale includes five grades of disability: from 0 to 5: 0 - no symptoms, 5 - gross disability; bedridden, fecal and urinary incontinence, need for constant assistance by medical staff.
Time Frame: On 90th day of the treatment.
Population: The number of completed cases (non-missing data) is indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 114 | 107
Participants | 57 | 53
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Test for comparison percentage of patients with no significant disabilities after 90 days of treatment; Test type: Superiority; p = 0.89, Fisher Exact

4. Secondary Outcome: Therapeutic and Side Effects, Efficacy Index.
Description: According to Clinical Global Impression Efficacy Index (CGI-EI).CGI-EI is filled out by an investigator. It is necessary to indicate the level of efficacy of the therapy and the grade of safety of the therapy and circle the index values at the intersection of the selected lines. Evaluation of the response to treatment should take into account both therapeutic efficacy and treatment-related side effects. Side effects score varies from 1 to 4 (lower is better). Therapeutic effect score varies from 1 to 4 (higher is better). The efficacy index is "Therapeutic effect score" divided by "Side effects score", so efficacy index varies from 0.25 to 4 (higher is better).
Time Frame: On 90th day of the treatment period.
Population: The number of completed cases (non-missing data) is indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 113 | 107
score on a scale
  Therapeutic effect | 3.3 (0.6) | 3.1 (0.7)
  Side effects | 1.2 (0.4) | 1.2 (0.5)
  Efficiency index | 3.0 (0.8) | 2.8 (0.9)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Therapeutic effect score comparison on 90th day of treatment; Test type: Superiority; p = 0.067, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: MMH-MAP vs Placebo; Side effects score comparison on 90th day of treatment; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: MMH-MAP vs Placebo; Efficacy index score comparison on 90th day of treatment; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Presence of Adverse Events (AEs).
Description: Based on medical records. Outcome measure represents the amount of participants having at least one adverse event on record.
Time Frame: For 90 days of the treatment period.
Measure: Number; unit: participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 123 | 122
participants | 32 | 28
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; The percentage of participants having at least one adverse event were compared; Test type: Superiority; p = 0.656, Fisher Exact

6. Secondary Outcome: Percentage of Patients With Complication of Cerebral Infarction.
Description: Based on medical records. The sequelae of cerebral infarction (severe infections - hospital-acquired pneumonia, uroinfection; deep venous thrombosis, PATE; epileptic episodes).
Time Frame: For 90 days of the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 122 | 119
Participants | 2 | 2
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Test type: Superiority; p = 1, Fisher Exact

7. Secondary Outcome: Death Rate.
Description: Based on medical records. Frequency of all-cause mortality outcomes.
Time Frame: For 90 days of the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 122 | 119
Participants | 0 | 0

8. Secondary Outcome: Changes in Vital Signs (Pulse Rate (Heart Rate)).
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: Visit 1 (day 1), Visit 2 (day 12), and Visit 4 (day 90).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 123 | 122
beats per minute
  Visit 1 (day 1) | 74.0 (7.6) | 73.5 (7.6)
  Visit 2 (day 12) | 71.3 (5.4) | 71.3 (6.3)
  Visit 4 (day 90) | 72.3 (6.1) | 71.4 (5.4)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Analysis of variance (ANOVA) for repeated measures has been used. Factors are "Treatment", "Visit" and interaction "Treatment-Visit". Significance of interaction as a factor representing difference in outcome value dynamics has been tested; Test type: Superiority; p = 0.96, ANOVA; P-value for interaction between factors "Treatment" and "Visit" is demonstrated

9. Secondary Outcome: Changes in Vital Signs (Respiration Rate (Breathing Rate)).
Description: Based on medical records. Vital signs will be measured in a medical setting.
Time Frame: Visit 1 (day 1), Visit 2 (day 12), and Visit 4 (day 90)
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 123 | 122
breaths per minute
  Visit 1 (day 1) | 16.8 (1.0) | 16.8 (0.9)
  Visit 2 (day 12) | 16.7 (1.0) | 16.7 (0.9)
  Visit 4 (day 90) | 16.8 (1.1) | 16.8 (1.0)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.96, ANOVA; P-value for interaction between factors "Treatment" and "Visit" is demonstrated

10. Secondary Outcome: Changes in Vital Signs (Blood Pressure).
Description: Based on medical records. Vital signs are measured in a medical setting. Systolic blood pressure (SBP) and diastolic blood pressure (DBP) are presented.
Time Frame: Visit 1 (day 1), Visit 2 (day 12), and Visit 4 (day 90).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 123 | 122
mmHg
  SBP/Visit 1 (day 1) | 139 (12.6) | 139.0 (11.2)
  SBP/Visit 2 (day 12) | 129 (8.3) | 130 (7.5)
  SBP/Visit 4 (day 90) | 129 (7.7) | 130 (7.8)
  DBP/Visit 1 (day 1) | 82.9 (7.0) | 83.5 (7.0)
  DBP/Visit 2 (day 12) | 80.0 (5.5) | 80.6 (5.7)
  DBP/Visit 4 (day 90) | 80.2 (5.3) | 80.0 (6.2)
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Systolic blood pressure. Analysis of varience (ANOVA) for repeated measures has been used. Factors are "Treatment", "Visit" and interaction "Treatment-Visit". Significance of interaction as a factor representing difference in outcome value dynamics has been tested; Test type: Superiority; p = 0.438, ANOVA; P-value for interaction between factors "Treatment" and "Visit" is demonstrated
Statistical Analysis 2: Comparison: MMH-MAP vs Placebo; Diastolic blood pressure. Analysis of variance (ANOVA) for repeated measures has been used. Factors are "Treatment", "Visit" and interaction "Treatment-Visit". Significance of interaction as a factor representing difference in outcome value dynamics has been tested; Test type: Superiority; p = 0.56, ANOVA; P-value for interaction between factors "Treatment" and "Visit" is demonstrated

11. Secondary Outcome: Percentage of Patients With Clinically Significant Abnormal Laboratory Data.
Description: Based on medical records. Laboratory tests include the following parameters (absolute and relative values): hematology, biochemistry and urinalysis. Laboratory tests will be made by central laboratory. Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L); greater than or equal to (>=)185 g/L; decreased from baseline (DFB) >=20 g/L Hematocrit: <=0.37 volume/volume (v/v); >=0.55 v/v Erythrocytes: >=6 Tera/L Leukocytes: >=16.0 Giga/L Neutrophils: <1.0 Giga/L (B); Lymphocytes: greater than (>) 4.0 Giga/L Monocytes: >0.7 Giga/L Basophils: >0.1 Giga/L Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L) Sodium: <=129 millimoles (mmol)/L; >=160 mmol/L Potassium: <3 mmol/L; >=5.5 mmol/L Alanine Aminotransferase (ALT): >3 ULN Aspartate aminotransferase (AST): >3 ULN Alkaline phosphatase: >1.5 ULN Bilirubin: >1.5 ULN Creatinine: >=150 micromoles per liter (mcmol/L); >=30% change from baseline.
Time Frame: On baseline and on 90th day of the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 123 | 122
Participants
  Baseline | 19 | 16
  On 90th day of the treatment | 2 | 1
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Comparison at the baseline; Test type: Superiority; p = 0.72, Fisher Exact
Statistical Analysis 2: Comparison: MMH-MAP vs Placebo; Comparison on 90th day of treatment; Test type: Superiority; p = 1, Fisher Exact

12. Secondary Outcome: Percentage of Patients With Recurring Cerebral Infarction.
Description: The percentage of patients with recurrent cerebral infarction for 90 days of the treatment period is estimated from medical records.
Time Frame: For 90 days of the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-MAP | Placebo
Number analyzed (Participants) | 122 | 119
Participants | 2 | 1
Statistical Analysis 1: Comparison: MMH-MAP vs Placebo; Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: Registration of AEs begins after taking the first dose of the study drug, continues throughout the entire period of study therapy - 90 days, as well as for 24 hours after the last dose of the study drug.
Arm/Group | MMH-MAP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/122
Serious Adverse Events (participants affected / at risk) | 4/123 | 4/122
Other Adverse Events (participants affected / at risk) | 32/123 | 28/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-MAP (N=123) | Placebo (N=122)
Recurrent stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Nosocomial pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hematoma as a complication of the procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Decompensated diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-MAP (N=123) | Placebo (N=122)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Discomfort in the epigastric region (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Coronavirus infection COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Abnormal renal ultrasound (Investigations) | 1 (1) | 0 (0)
Increased blood pressure (Investigations) | 3 (3) | 4 (4)
Increased blood glucose (Investigations) | 2 (2) | 0 (0)
Increased body temperature (Investigations) | 0 (0) | 1 (1)
Lower blood pressure (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic decompensation of diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron-deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemorrhagic transformation after stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Acute cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Wax plug (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 3 (3)
Peripheral edema (General disorders) | 0 (0) | 2 (2)
Deterioration of condition (General disorders) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder associated with general somatic (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hematoma after procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT04295681/Prot_SAP_000.pdf